CLINICAL TRIAL: NCT06660030
Title: Factors Influencing Tamoxifen Adherence in Women With Breast Cancer Receiving Tamoxifen in Botswana.
Acronym: TAM
Status: Terminated | Type: Observational
Why Stopped: Lack of funds
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 855696
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Approximately 4 ml of blood will be drawn from consenting patients following questionnaire administration in EDTA ( this is an anticoagulant to collect whole blood in tubes ) tubes. Blood will be immediately centrifuged after collection, and plasma and buffy coat stored for drug/metabolites detection/quantification, and DNA analysis, respectively.
  DNA extraction technique:( this is a DNA extraction kit) QIAamp DNA Mini Kits (Qiagen, Hilden, Germany) kits will be used for whole genomic DNA, according to the manufacture's instructions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Botswana is an ideal location to investigate tamoxifen adherence for numerous reasons. First, in contrast to many other countries in SSA, tamoxifen is affordable and widely available to women with ER+ breast cancer in Botswana. There is also a sufficiently high prevalence of WLW HIV and breast cancer in Botswana to provide adequate power for the proposed study. Lastly, there is a well-developed medical and scientific infrastructure, both from the clinical and laboratory perspective, to allow for successful completion of this proposed study

DETAILED DESCRIPTION:
Breast cancer (BC) is the second-most common cancer in women in sub-Saharan Africa (SSA) (Black 2019, Trimble 2017). Tamoxifen forms a cornerstone for treatment of ER+ breast cancer and daily use after initial medical, surgical, and/or radiation therapy decreases the annual odds of recurrence and death by 39% and 31% respectively (EBCTCG 2005). Despite the proven benefits of tamoxifen, non-adherence is common. Previous reports have indicated that 31-50% of women do not adhere to prescribed treatment regimens (Lash 2006, Lambert 2018, Peddie 2021). The reasons for non-adherence are broad and not fully understood but are thought to be influenced by numerous factors including medication side-effects, beliefs about cancer, and social support framework (Clancy 2020). Data is extremely limited concerning the adherence rates to tamoxifen therapy in Africa.

The metabolism of tamoxifen is complex. It is metabolized to its effector/active metabolites via the cytochrome P450 (CYP) enzyme system, principally CYP2D6 with CYP2B6 playing a lesser, but important role (Nthontho Keneuoe Cecilia 2022). The CYP2D6 gene is highly variable but four principal drug metabolizer phenotypes have been identified: poor, intermediate, extensive, and ultra-rapid metabolizers (Nthontho KC 2022). Reduced speed of tamoxifen metabolism in poor metabolizers has been associated with higher risk of treatment failure, due to increased drug level in vivo and subsequent increased tamoxifen related side effects (Nardin 2020). However, to date, these various phenotypes have not been evaluated in an African population, so it is unclear to what extent these phenotypes effect tamoxifen adherence in SSA.

A unique aspect among the breast cancer population in Botswana is that a large portion of these women are also living with HIV. Studies have shown that the prevalence of HIV in the general population is up to 17.6% (Bhatia 2019). Little is known how antiretroviral medications effect tamoxifen adherence. One particular Anti Retroviral Therapy (ART) medication, efavirenz (EFV), a non-nucleoside reverse transcriptase inhibitor and potent CYP-inducer is used by a large portion of WLW HIV in SSA (Maseng 2022). EFV has been shown in vitro to increase estrogen expression both by inducing growth in ER-positive breast cancer cells lines (Sikora 2010) and clinically due to the development of gynecomastia seen in male patients (Osman 2020). It remains unclear, however, if and to what extent the combined administration of tamoxifen and efavirenz contributes to reduced tamoxifen adherence.

ELIGIBILITY:
Inclusion Criteria.

* All women over the age of 18, taking (or have taken) tamoxifen for treatment of ER+ breast cancer and being HIV positive
* All women over the age of 18, taking (or have taken) tamoxifen for treatment of ER+ breast cancer and being HIV negative

Exclusion Criteria:

* Males
* Women with ER negative breast cancer
* Women under 18 years of age at time of study administration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with breast cancer
Study Population: Patients will include females with ER+ breast cancer who are >18 years of age. The study population will include both women living with and without HIV.
  Patients offered questionnaires and blood draws will only include women treated as outpatients and be of sufficient mental capacity to personally consent to the study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Primary outcome | 12 months
  Reduced tamoxifen adherence, measured as reduced intake of pills number will be seen in women with reduced quality of EORTC QLQ( Cancer core quality of life questionnare acronym Q-C30 life scores, increased medication side effects, and/or increased barriers to medical care.
  Women living with (WLW) HIV taking tamoxifen will be less adherent to tamoxifen therapy due to the higher likelihood of medication side effects

SECONDARY OUTCOMES:
Secondary outcome | 12 months
  Women identified as poor metabolizers will have higher tamoxifen and metabolite plasma concentrations (measured as mg/ml).

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Marina Hospital, Gaborone, Botswana